



## A BEHAVIORAL INTERVENTION WITH FOSTER FAMILIES

NCT Number: In progress of registering

Date of Original Document: January 4, 2022

**Consent Form** 

HSPP Use Only: Consent Script Non-Funded or Internally-Funded v2021-09-02





University of Arizona
Consent and/or Parental Permission to Participate in Research

Study Title: Effects of a Behavioral Intervention with Foster Families

## **Principal Investigator:**

References to "you" and "your" throughout this document refer to both you and your child(ren).

You are being asked to participate in a research study. Your participation in this research study is voluntary and you do not have to participate. This document contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to ask questions before making your decision on whether to participate.

This study will be investigating an online family learning video and activities meant to help prepare and strengthen your family as you take in foster children with special needs. It is self-paced and includes 4 videos with activities that you will be asked to complete over a 1-month period.

Your family will be randomly assigned by a statistician to a control or intervention group. The control group will not participate in the intervention during the study period. If your family is randomized to the control group, you will only be asked to fill out the survey at the beginning of one month and then again at the end of the month. Should you choose to participate in the salivary cortisol collection (saliva by passive drool), you will be asked to collect saliva at 3 separate times: at the beginning of the study, one month later, and again another month later.

Involvement in the intervention group study includes:

- 1. Answering a 15-minute survey online before, after, and then 1-month after finishing the videos
- 2. Watching all 4 videos/learning modules with activities.
- 3. Including at least one child in your home (ideally, the child that is closest in age to your foster child) in the intervention (videos and activities).
- 4. Optional (not all families will participate passive collection of saliva samples on 3 separate intervals for 3 days each (before study, after the intervention, and 1 month after the intervention) of you and one child for whom you are the legal guardian.

Your child (children) will be asked to view mini videos with you and do a family-building activity 4 times during the study. Benefits include that you will be able to participate in an adapted program from the Karyn Purvis Institute of Childhood Development that is meant to improve family functioning and attachment within foster families.



Additionally, you will be helping researchers develop tools to help foster families and children in foster care to have positive outcomes.

There are no expected risks to you because of participating in this study. Your identity and family information will be kept confidential. Expected time commitment is 15 minutes for 3 surveys. If you are in the intervention group you will have four separate videos/activities that take approximately 30 minutes each. These will be spaced out between 4 weeks (30 minutes each week for a total of 4 times). If you are part of the saliva collection group, you will collect saliva samples for you and one child on three different time points (before the study, after the intervention, and one month later) on three separate days at each time point. Saliva collection occurs over three separate days and is done at waking, 30 minutes after waking, and at bedtime on each of those days for a total of 27 samples per participant. Saliva is stored in containers provided to you and placed in your freezer. Once collection of samples is completed, you will place the samples in the prepaid shipping container, which a courier will pick up. Time to collect saliva, label, and store sample takes less than 5 minutes each time (average time is 2 minutes for each saliva sample collected).

The control groups complete the 3 surveys (15 minutes each). Some of the control group participants will participate in saliva collection as well (before the study, when intervention group completes the intervention, and one month later). There are no other costs to participating in the study and all supplies and shipping of samples will be prepaid by the study group.

You will be compensated 3 separate times: upon completion of the initial survey (\$25), after the intervention (\$25), and again after the final saliva collection (\$25) for up to \$75 total.

Compensation for participation in a research study is considered taxable income for you. If your compensation for this research study or a combination of research studies is \$600 or more in a calendar year (January to December), you will receive an IRS Form 1099 to report on your taxes. Please note, if you are an employee of UArizona, any compensation from a research study is considerable taxable income.

For any compensation or reimbursement you receive, we are required to obtain identifiable information such as your name and address.

Your participation is voluntary. You do not need to participate in this study. If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with The University of Arizona. If you are a student or employee at the University of Arizona, your decision will not affect your grades or employment status.



Consent Version: 12/27/2021

Page 4 of 5

Your name will not be used in any report. Identifiable research data will be encrypted, and password protected.

Your responses will be assigned a code number. The list connecting your name to this code will be kept in an encrypted and password protected file. Only the research team will have access to the file. When the study is completed and the data have been analyzed, the list will be destroyed.

Because of the nature of the data, it may be possible to deduce your identity; however, there will be no attempt to do so, and your data will be reported in a way that will not identify you.

De-identified data from this study may be used for future research or shared with another researcher for future research studies without additional consent.

The information that you provide in the study will be handled confidentially. However, there may be circumstances where this information must be released or shared as required by law. The University of Arizona Institutional Review Board may review the research records for monitoring purposes.

| For questions, concerns, or c | omplaints about the study you m | ay contact |
|---|---|---|
| concerns or complaints with the Human Subjects Protection | hts as a participant in this study o<br>someone who is not part of the r<br>on Program Director at 520-626-8<br>/compliance/human-subjects-pro | esearch team, you may contact<br>3630 or online at |
| By taking part in our online so purposes. | urvey, you are allowing your resp | onses to be used for research |
| | esearch team member to contact<br>ated content. Agree Disagre | |
| participate in a research studentswered to my satisfaction. | I voluntarily agree to participate | ask questions and have had them in this study. |
| i am not giving up any legal r | ights by signing this form. I will b | e given a copy of this form. |
| Printed name of subject | Signature of subject | Date |



Name of child

Consent Version: 12/27/2021 Page 5 of 5

| Name of child |
|---------------|
| Name of child |
| Name of child |

HSPP Use Only: Consent Script Non-Funded or Internally-Funded v2021-09-02